CLINICAL TRIAL: NCT00544050
Title: An Open-Label, Single Dose, Pharmacokinetic Study of 20 mg/kg of Levetiracetam Oral Solution in Epileptic Pediatric Subjects Ranging in Age From 1 Month to Less Than 4 Years Old
Brief Title: Pharmacokinetic Study of Levetiracetam in Epileptic Pediatric Subjects Ranging in Age From 1 Month to Less Than 4 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01052
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2009-09

CONDITIONS: Epilepsy
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
The primary purpose of this study was to document the pharmacokinetic parameters of both levetiracetam and its metabolite, ucb L057, after a single dose of 20 mg/kg of levetiracetam in epileptic pediatric subjects, aged 1 month to less than 4 years.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 1 month and less than 4 years
* diagnosis of any type of epilepsy
* at least 5 kg body weight
* using no more than two antieplieptic drugs

Exclusion Criteria:

* a treatable seizure etiology
* epilepsy secondary to a progressive cerebral disease or any other progressively neurodegenerative disease
* history of status epilepticus during the 2 weeks prior to the Selection Visit
* history of or the presence of pseudoseizures
* epilepsy surgery within one year prior to the Selection Visit
* on a ketogenic diet
* taking felbamate at the Selection Visit

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2002-09; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
PK parameters of both levetiracetam and its metabolite, ucb L057, after a single dose of 20 mg/kg levetiracetam.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Background] Glauser TA, Mitchell WG, Weinstock A, Bebin M, Chen D, Coupez R, Stockis A, Lu ZS. Pharmacokinetics of levetiracetam in infants and young children with epilepsy. Epilepsia. 2007 Jun;48(6):1117-22. doi: 10.1111/j.1528-1167.2007.01090.x. Epub 2007 Apr 18. PMID 17442002